CLINICAL TRIAL: NCT00110214
Title: A Randomized Double-Blinded Placebo Controlled Phase III Trial Comparing Doctaxel and Prednisone With and Without Bevacizumab (IND #7921, NSC #704865) in Men With Hormone Refractory Prostate Cancer
Brief Title: Docetaxel and Prednisone With or Without Bevacizumab in Treating Patients With Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02814; NCI-2012-02814 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000427290; CALGB-90401 (Other: Cancer and Leukemia Group B); CALGB-90401 (Other: CTEP); P30CA014236 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2005-05-04; First posted 2005-05-05 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2012-12

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Experimental): Patients receive docetaxel IV over 1 hour and placebo IV over 30-90 minutes on day 1. Patients also receive oral prednisone once daily on days 1-21.
  Interventions: Drug: docetaxel; Other: placebo; Drug: prednisone; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive docetaxel and prednisone as in arm I. Patients also receive bevacizumab IV over 30-90 minutes on day 1.
  Interventions: Drug: docetaxel; Drug: prednisone; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Other: placebo — Given IV
  Other Names: PLCB
  Arms: Arm I
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm II
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase III trial is studying docetaxel, prednisone, and bevacizumab to see how well they work compared to docetaxel and prednisone in treating patients with prostate cancer that did not respond to hormone therapy. Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether docetaxel, prednisone, and bevacizumab are more effective than docetaxel and prednisone in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of bevacizumab to docetaxel and prednisone increases overall survival compared to docetaxel and prednisone alone in patients with HRPC.

SECONDARY OBJECTIVES:

I. To compare the progression-free survival of these two regimens in patients with HRPC.

II. To compare the two regimens on the proportion of patients who experience a 50% post-therapy PSA decline from baseline.

III. To compare the two regimens with respect to the proportion of patients who experience grade 3 or higher toxicities.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to predicted 24-month survival probability (< 10% vs 10-29.9% vs ≥ 30%), age (< 65 years vs ≥ 65 years), and prior history of arterial events (i.e., cardiac ischemia/infarction, CNS cerebrovascular ischemia, peripheral arterial ischemia, or CNS hemorrhage) (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive docetaxel IV over 1 hour and placebo IV over 30-90 minutes on day 1. Patients also receive oral prednisone once daily on days 1-21.

ARM II: Patients receive docetaxel and prednisone as in arm I. Patients also receive bevacizumab IV over 30-90 minutes on day 1.

In both arms, courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented adenocarcinoma of the prostate with progressive systemic (clinically metastatic disease documented on bone, CT or MRI scan) disease despite castrate levels of testosterone due to orchiectomy or LHRH agonist; castrate levels of testosterone must be maintained
* All eligible patients must have a Gleason sum based on biopsy or TURP at the time of registration
* At the time of enrollment, patients must have evidence of progressive metastatic disease, either:

  * Measurable disease with any level of serum PSA OR
  * Non-measurable disease with PSA ≥ 5 ng/ml; patients with PSA ≥ 5 ng/ml only and no other radiographic evidence of metastatic prostate cancer are not eligible
* Definition of Measurable Disease/Target Lesions:

  * Any lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques: 1) physical exam for clinically palpable lymph nodes and superficial skin lesions, 2) chest X-ray for clearly defined lung lesions surrounded by aerated lung OR those lesions measured as ≥ 10 mm with a spiral CT or MRI scan
  * Measurable lesions (up to a maximum of 10 in number) representative of all organs involved to be identified as target lesions; the sum of the longest diameters (LD) for all target lesions will be calculated and reported as baseline sum LD

    * If measurable disease is confined to a solitary lesion and is not consistent with prostate cancer, then its neoplastic nature must be confirmed by histology
    * Ultrasound may not be used to measure tumor lesions that are not easily accessible clinically
* Definition of Non-measurable Disease/Non-target Lesions:

  * Non-target lesions include all other lesions not included in above, including small lesions with longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan and truly non-measurable lesions, which include:

    * Bone lesions
    * Pleural or pericardial effusions, ascites
    * CNS lesions, leptomeningeal disease
    * Irradiated lesions, unless progression documented after RT
* Patients must have demonstrated evidence of progressive disease since the most recent change in therapy; progressive disease is defined as any one of the following (measurable disease, bone scan, or PSA progression):

  * Measurable Disease Progression: Objective evidence of increase > 20% in the sum of the longest diameters (LD) of target lesions from the time of maximal regression or the appearance of one or more new lesions
  * Bone Scan Progression: Appearance of one or more new lesions on bone scan attributable to prostate cancer along with a PSA ≥ 5 ng/ml will constitute progression
  * PSA Progression: An elevated PSA (≥ 5 ng/mL) which has risen serially on at least two occasions after the discontinuation of antiandrogen therapy, each at least one week apart; if the confirmatory PSA (#3) value is less than screening PSA (#2) value, then an additional test for rising PSA (#4) will be required to document progression

    * The reference PSA value (#1) must be measured at the time of the discontinuation of antiandrogen therapy; and at least 2 PSA measurements must be made following the end of antiandrogen therapy and prior to registration
    * (For the purposes of the nomogram calculator, the last PSA value recorded prior to the initiation of treatment will be considered the baseline PSA)
* Progression despite standard androgen deprivation therapy (i.e., LHRH agonist and/or orchiectomy)
* All antiandrogens (e.g., flutamide, megestrol acetate [even if taken for hot flashes], bicalutamide and nilutamide) of any dose must be discontinued at least 4 weeks prior to registration; if improvement following antiandrogen withdrawal is noted, progression must be established using the criteria above

  * Primary testicular androgen suppression (e.g., with an LHRH agonist) should not be discontinued
* At least 4 weeks since any other hormonal therapy, including ketoconazole and aminoglutethimide; the only exception to this time frame is that 5α-reductase inhibitors (e.g., finasteride, dutasteride) may be discontinued any time prior to registration
* No prior cytotoxic chemotherapy, including estramustine or suramin
* No prior anti-angiogenesis agents, including thalidomide and bevacizumab
* ≥ 4 weeks since major surgery and fully recovered
* ≥ 4 weeks since any prior radiation (including palliative) and fully recovered
* ≥ 8 weeks since the last dose of Strontium-89 or Samarium
* Patients receiving a bisphosphonate must be on a stable dose and must have started the bisphosphonate ≥ 4 weeks prior to initiating protocol treatment. Patients do not have to be on a bisphosphonate to qualify for the study; patients may initiate bisphosphonate therapy after completion of Cycle 1, if clinically indicated

  * Patients enrolled on CALGB 90202 who have documented disease progression and have received at least 4 weeks of open label zoledronic acid treatment, are eligible for this study.
* No known brain metastases (brain imaging (MRI/CT) is not required)
* No current congestive heart failure (New York Heart Association Class II, III or IV)
* Patients with history of hypertension must be well controlled (< 160/90) on a regimen of anti-hypertensive therapy
* Patients on full-dose anticoagulants must be on a stable dose of warfarin and have an in-range INR (usually between 2 and 3) or be on a stable dose of LMW heparin; patients receiving anti-platelet agents are also eligible; in addition, patients who are on daily prophylactic aspirin or anticoagulation for atrial fibrillation are eligible
* No significant history of bleeding events or GI perforation

  * Patients with a history of significant bleeding episodes (e.g., hemoptysis, upper or lower GI bleeding) within 6 months of registration are not eligible
  * Patients with a history of GI perforation within 12 months of registration are not eligible.
* No recent (within 12 months) arterial thrombotic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina or angina requiring surgical or medical intervention in the past 12 months, or myocardial infarction (MI); patients with clinically significant peripheral artery disease (i.e., claudication on less than one block) or any other arterial thrombotic event are also ineligible
* No serious or non-healing wound, ulcer or bone fracture
* No peripheral neuropathy ≥ grade 2
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies are not eligible
* PC-Spes, Saw Palmetto, and St. John's Wort must be discontinued before registration; the discontinuation of other herbal medications and food supplements is strongly encouraged; patients may continue on daily vitamins and calcium supplements
* ECOG performance status: 0-2
* ANC ≥ 1500/μL
* Platelet count ≥ 100,000/μL
* Creatinine ≤ 1.5 x upper limits of normal
* Bilirubin ≤ 1.5 x upper limits of normal

  * For patients with Gilbert's Disease, ≤ 2.5 X ULN is allowed
* AST ≤ 1.5 x upper limits of normal
* PSA ≥ 5 ng/mL (if non-measurable disease)
* Urine protein to creatinine ratio < 1.0

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2005-04; Primary Completion 2010-03 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kelly, Principal Investigator — Cancer and Leukemia Group B
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Cancer and Leukemia Group B, Chicago, Illinois

REFERENCES:
- [Derived] Quintanilha JCF, Kelly WK, Innocenti F. Contribution of plasma levels of VEGF-A and angiopoietin-2 in addition to a genetic variant in KCNAB1 to predict the risk of bevacizumab-induced hypertension. Pharmacogenomics J. 2024 Jul 12;24(4):22. doi: 10.1038/s41397-024-00342-1. PMID 38992025
- [Derived] Quintanilha JCF, Wang J, Sibley AB, Jiang C, Etheridge AS, Shen F, Jiang G, Mulkey F, Patel JN, Hertz DL, Dees EC, McLeod HL, Bertagnolli M, Rugo H, Kindler HL, Kelly WK, Ratain MJ, Kroetz DL, Owzar K, Schneider BP, Lin D, Innocenti F. Bevacizumab-induced hypertension and proteinuria: a genome-wide study of more than 1000 patients. Br J Cancer. 2022 Feb;126(2):265-274. doi: 10.1038/s41416-021-01557-w. Epub 2021 Oct 6. PMID 34616010
- [Derived] Quintanilha JCF, Liu Y, Etheridge AS, Yazdani A, Kindler HL, Kelly WK, Nixon AB, Innocenti F. Plasma levels of angiopoietin-2, VEGF-A, and VCAM-1 as markers of bevacizumab-induced hypertension: CALGB 80303 and 90401 (Alliance). Angiogenesis. 2022 Feb;25(1):47-55. doi: 10.1007/s10456-021-09799-1. Epub 2021 May 24. PMID 34028627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2005 and December 2007, 1,050 participants were recruited and randomized
Groups:
- Docetaxel + Placebo: Standard treatment Docetaxel: 75 mg/m2 by IV over 1 hour for 21 days, Prednisone: 5mg orally twice per day Placebo
- Docetaxel + Bevacizumab: Std Tx + monoclonal antibody therapy Docetaxel: 75 mg/m2 by IV over 1 hour for 21 days, Prednisone: 5mg orally twice per day Bevacizumab: 15 mg/kg IV every 3 weeks
Period: Overall Study
Arm/Group | Docetaxel + Placebo | Docetaxel + Bevacizumab
Started | 526 | 524
Completed | 17 | 21
Not Completed | 509 | 503
Not completed — Never started treatment | 21 | 20
Not completed — Disease progression or death | 260 | 151
Not completed — Adverse Event | 115 | 192
Not completed — Refused further treatment | 52 | 65
Not completed — Other (not specified) | 61 | 75

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel + Placebo | Docetaxel + Bevacizumab | Total
Number analyzed (Participants) | 526 | 524 | 1050
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.3 [62.4 to 75.6] | 68.8 [63.0 to 74.4] | 69.0 [62.7 to 75.2]
Age, Customized [Number; unit: participants]
  < 65 years | 174 | 179 | 353
  >=65 years | 352 | 345 | 697
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 526 | 524 | 1050
Region of Enrollment [Number; unit: participants]
  United States | 526 | 524 | 1050
24-month predicted survival probability [Number; unit: participants]
  <10% | 95 | 94 | 189
  10-29.9% | 184 | 183 | 367
  >=30% | 247 | 247 | 494
Prior history of arterial events [Number; unit: participants]
  Yes | 42 | 37 | 79
  No | 484 | 487 | 971

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall Survival (OS) was measured from the date of randomization to date of death due to any cause. OS was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Placebo | Docetaxel + Bevacizumab
Number analyzed (Participants) | 526 | 524
months | 21.5 [20.0 to 23.0] | 22.6 [21.1 to 24.5]
Statistical Analysis 1: Comparison: Docetaxel + Placebo vs Docetaxel + Bevacizumab; Test type: Non-Inferiority or Equivalence — Superiority and futility analyses were conducted for the OS end point. The Lan-Demets analog of the Emerson-Fleming sequential boundary was used to maintain the overall significance level of alpha=0.05 while conducting interim analyses on OS. The final analysis was performed when 748 deaths had been observed. An intention-to-treat approach was used in the analysis for all the clinical end points with the exception of toxicity; p = 0.181, Log Rank — The primary analysis was adjusted for the stratification factors (24-mo survival probability as predicted by a validated nomogram (<10%,10%-29.9%,>=30%), age (<65, >=65 years) and prior history of arterial events (yes, no)); Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.7 to 1.05]

2. Secondary Outcome: Proportion of Participants Who Experienced at Least a 50% Post-therapy PSA (Prostate-Specific Antigen) Decline
Description: PSA decline will be reported on all patients and will be defined as a decrease in PSA value by >= 50% for two successive evaluations at least 4 weeks apart. The reference PSA value for these declines should be measured within 2 weeks before starting therapy.
Time Frame: Duration of study (up to 5 years)
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel + Placebo | Docetaxel + Bevacizumab
Number analyzed (Participants) | 526 | 524
percentage of participants | 57.9 | 69.5
Statistical Analysis 1: Comparison: Docetaxel + Placebo vs Docetaxel + Bevacizumab; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the data of randomization to date of progression or death due to any cause, whichever occurs first. PFS was estimated using the Kaplan Meier method.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Duration of study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Placebo | Docetaxel + Bevacizumab
Number analyzed (Participants) | 526 | 524
months | 7.5 [6.8 to 8.0] | 9.9 [9.0 to 10.6]
Statistical Analysis 1: Comparison: Docetaxel + Placebo vs Docetaxel + Bevacizumab; Test type: Superiority or Other; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.71 to 0.91]

4. Secondary Outcome: Proportion of Participants Who Experience (Maximum) Grade 3 or Higher Toxicities
Description: The National Cancer Institute (NCI) Criteria for Adverse Events(CTCAE) Version 3.0 was used to evaluate toxicity. These events were considered at least possibly related to treatment.
  Grade 1: mild; Grade 2: moderate; Grade 3: Severe; Grade 4: Life Threatening; Grade 5: Death
Time Frame: During treatment (up to 2 years)
Population: Participants who did not received allocated intervention were excluded from toxicity analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel + Placebo | Docetaxel + Bevacizumab
Number analyzed (Participants) | 505 | 504
percentage of participants | 56.2 | 75.4

ADVERSE EVENTS:
Description: Participants who did not received allocated intervention were excluded from toxicity analysis
Arm/Group | Docetaxel + Placebo | Docetaxel + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 237/505 | 178/504
Other Adverse Events (participants affected / at risk) | 420/505 | 363/504
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + Placebo (N=505) | Docetaxel + Bevacizumab (N=504)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (26) | 19 (21)
Hemoglobin (Blood and lymphatic system disorders) | 17 (19) | 14 (15)
Lymphatics - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac General - Other (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 12 (12) | 4 (4)
Cardiopulmonary arrest cause unknown (non-fatal) (Cardiac disorders) | 1 (1) | 0 (0)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 0 (0) | 2 (3)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 2 (3)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 8 (8) | 10 (11)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Thyroid function high (hyperthyroidism thyrotoxicosis) (Endocrine disorders) | 0 (0) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1)
Watery eye (epiphora tearing) (Eye disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 9 (10)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fistula, GI (Gastrointestinal disorders) | 6 (6) | 2 (3)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 4 (4) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI (Gastrointestinal disorders) | 38 (42) | 18 (19)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 8 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 16 (18) | 5 (5)
Obstruction GI (Gastrointestinal disorders) | 2 (2) | 1 (1)
Perforation, GI (Gastrointestinal disorders) | 19 (20) | 3 (3)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcer GI (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ulcer, GI (Gastrointestinal disorders) | 4 (5) | 1 (2)
Vomiting (Gastrointestinal disorders) | 10 (10) | 4 (4)
Death not associated with CTCAE term (General disorders) | 10 (10) | 10 (10)
Edema: limb (General disorders) | 1 (1) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 39 (46) | 22 (27)
Fever (General disorders) | 43 (47) | 32 (35)
Injection site reaction/extravasation changes (General disorders) | 1 (1) | 0 (0)
Pain - Other (General disorders) | 5 (6) | 3 (3)
Rigors/chills (General disorders) | 13 (15) | 17 (20)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Necrosis GI (Hepatobiliary disorders) | 1 (1) | 0 (0)
Necrosis, GI (Hepatobiliary disorders) | 1 (1) | 0 (0)
Obstruction, GI (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (3) | 3 (3)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 3 (3) | 2 (3)
Infection (Infections and infestations) | 35 (41) | 27 (30)
Infection - Other (Infections and infestations) | 14 (14) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 18 (19) | 11 (15)
Infection with unknown ANC (Infections and infestations) | 13 (13) | 3 (3)
Infection without neutropenia (Infections and infestations) | 2 (2) | 0 (0)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 2 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (2)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication non-infectious (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I (cTnI) (Investigations) | 4 (4) | 1 (1)
Cardiac troponin T (cTnT) (Investigations) | 1 (1) | 0 (0)
Coagulation - Other (Investigations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 2 (3) | 2 (2)
Fibrinogen (Investigations) | 1 (1) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Investigations) | 39 (48) | 25 (28)
Lymphopenia (Investigations) | 11 (14) | 11 (14)
Metabolic/Laboratory - Other (Investigations) | 0 (0) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 67 (79) | 46 (58)
Neutrophils/granulocytes (ANC/AGC) for BMT studies if specified in the protocol. (Investigations) | 0 (0) | 1 (1)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1) | 2 (2)
Platelets (Investigations) | 2 (3) | 0 (0)
Weight gain (Investigations) | 1 (3) | 0 (0)
Weight loss (Investigations) | 2 (2) | 0 (0)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 14 (15) | 5 (5)
Calcium serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (7) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 27 (32) | 14 (17)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 11 (12) | 6 (8)
Glucose serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4) | 5 (6)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 10 (10) | 6 (6)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 11 (11) | 3 (3)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 2 (2) | 3 (3)
CNS cerebrovascular ischemia (Nervous system disorders) | 5 (5) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 7 (8)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Hemorrhage CNS (Nervous system disorders) | 0 (0) | 2 (2)
Neurology - Other (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 5 (5) | 4 (6)
Neuropathy: sensory (Nervous system disorders) | 4 (4) | 7 (8)
Pain (Nervous system disorders) | 25 (27) | 19 (24)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 (3) | 2 (3)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 9 (10) | 7 (8)
Confusion (Psychiatric disorders) | 2 (2) | 5 (5)
Mood alteration (Psychiatric disorders) | 2 (2) | 0 (0)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Fistula, GU (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage GU (Renal and urinary disorders) | 6 (7) | 9 (10)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstruction, GU (Renal and urinary disorders) | 1 (1) | 5 (5)
Perforation GU (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 22 (26) | 19 (21)
Renal failure (Renal and urinary disorders) | 3 (4) | 5 (6)
Stricture/stenosis (including anastomotic), GU (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 3 (3) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 12 (13)
Hemorrhage pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 3 (3)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice changes/dysarthria (e.g. hoarseness loss or alteration in voice laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (8) | 10 (15)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (hives welts wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes/flushes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 24 (27) | 6 (9)
Hypotension (Vascular disorders) | 11 (11) | 6 (7)
Thrombosis/thrombus/embolism (Vascular disorders) | 17 (17) | 28 (31)
Vascular - Other (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + Placebo (N=505) | Docetaxel + Bevacizumab (N=504)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (15) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 12 (20) | 9 (11)
Hemolysis (e.g. immune hemolytic anemia drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphatics - Other (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac General - Other (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 4 (4) | 3 (3)
Edema (Cardiac disorders) | 0 (0) | 1 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (3) | 2 (2)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Otitis middle ear (non-infectious) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1) | 3 (8)
Watery eye (epiphora tearing) (Eye disorders) | 10 (23) | 2 (10)
Constipation (Gastrointestinal disorders) | 7 (8) | 2 (2)
Dental: periodontal disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 18 (19) | 7 (9)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (6) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fistula, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (2) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI (Gastrointestinal disorders) | 33 (46) | 13 (19)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus GI (functional obstruction of bowel i.e. neuroconstipation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incontinence anal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 6 (7) | 0 (0)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 12 (20) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (13) | 7 (7)
Perforation, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 2 (11) | 0 (0)
Ulcer, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (4)
Death not associated with CTCAE term (General disorders) | 1 (1) | 2 (2)
Edema: limb (General disorders) | 1 (1) | 5 (8)
Edema: trunk/genital (General disorders) | 0 (0) | 1 (5)
Extremity-lower (gait/walking) (General disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 90 (157) | 51 (80)
Fever (General disorders) | 77 (105) | 50 (64)
Pain - Other (General disorders) | 4 (4) | 6 (8)
Rigors/chills (General disorders) | 42 (73) | 33 (67)
Syndromes - Other (General disorders) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 20 (56) | 26 (47)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 29 (40) | 15 (18)
Infection - Other (Infections and infestations) | 12 (23) | 6 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 36 (61) | 21 (28)
Infection with unknown ANC (Infections and infestations) | 25 (33) | 10 (14)
Infection without neutropenia (Infections and infestations) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vessel injury-artery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 (6) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (3) | 2 (2)
Alkaline phosphatase (Investigations) | 12 (18) | 12 (29)
CD4 count (Investigations) | 1 (4) | 0 (0)
Cholesterol serum-high (hypercholesteremia) (Investigations) | 1 (4) | 0 (0)
Creatinine (Investigations) | 0 (0) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 2 (5) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 0 (0) | 3 (3)
Leukocytes (total WBC) (Investigations) | 56 (176) | 50 (113)
Lymphopenia (Investigations) | 18 (87) | 31 (90)
Metabolic/Laboratory - Other (Investigations) | 4 (12) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 110 (312) | 97 (252)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1) | 1 (1)
Platelets (Investigations) | 2 (6) | 0 (0)
Weight gain (Investigations) | 0 (0) | 2 (19)
Weight loss (Investigations) | 5 (10) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (15) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 14 (24) | 5 (7)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 48 (142) | 40 (82)
Magnesium serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (5) | 2 (2)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (6) | 1 (2)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9 (13) | 3 (5)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 7 (13) | 10 (11)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 2 (3) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 2 (2) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage CNS (Nervous system disorders) | 1 (2) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: cranial (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 9 (14) | 17 (32)
Neuropathy: sensory (Nervous system disorders) | 33 (50) | 33 (67)
Pain (Nervous system disorders) | 44 (64) | 34 (43)
Pyramidal tract dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 5 (6) | 5 (7)
Taste alteration (dysgeusia) (Nervous system disorders) | 3 (10) | 1 (1)
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Mood alteration (Psychiatric disorders) | 3 (6) | 1 (1)
Personality/behavioral (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder spasms (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Fistula, GU (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Hemorrhage GU (Renal and urinary disorders) | 2 (4) | 6 (8)
Incontinence, urinary (Renal and urinary disorders) | 3 (13) | 3 (4)
Obstruction, GU (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 89 (295) | 70 (174)
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 (1) | 0 (0)
Stricture/stenosis (including anastomotic), GU (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 4 (4)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 5 (12) | 4 (8)
Allergic rhinitis (including sneezing nasal stuffiness postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 7 (7)
Hemorrhage pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 153 (603) | 54 (123)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Voice changes/dysarthria (e.g. hoarseness loss or alteration in voice laryngitis) (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 7 (17) | 5 (12)
Nail changes (Skin and subcutaneous tissue disorders) | 8 (17) | 5 (7)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 69 (155) | 56 (119)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (11) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (hives welts wheals) (Skin and subcutaneous tissue disorders) | 10 (15) | 4 (8)
Dermal change lymphedema phlebolymphedema (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 (0) | 2 (2)
Hot flashes/flushes (Vascular disorders) | 4 (6) | 0 (0)
Hypertension (Vascular disorders) | 156 (568) | 82 (198)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 7 (12) | 20 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less